CLINICAL TRIAL: NCT05032079
Title: Pilot Study for the Cryoablation of Ductal Carcinoma In Situ: Subzero and Scorpion Trial
Brief Title: Subzero and Scorpion Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study Period Ended / Not Completed
Sponsor: Larkin Community Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCH-112020
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Ductal Carcinoma in Situ
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Procedure: cryoablation

INTERVENTIONS:
Procedure: cryoablation — single probe ultrasound guided cryoablation
  Other Names: cryosurgery

SUMMARY:
This is a prospective single-institution pilot study examining the feasibility of performing ultrasound-guided cryoablation to completely ablate breast ductal carcinoma in situ (DCIS). The study is designed such that patients meeting selection criteria will undergo cryoablation followed by surgical resection. The pathology of the surgical specimen will be used to determine the rate of complete tumor ablation. Standard adjuvant therapies otherwise remained unchanged.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18
2. Pre-registration core biopsy:

   Unifocal primary ductal carcinoma in situ (DCIS) or atypical ductal hyperplasia (ADH) bordering on DCIS or DCIS with microinvasion diagnosed by core needle biopsy. NOTE: Patients with lobular carcinoma, multifocal and/or multicentric ipsilateral breast cancer are NOT eligible. Patients with contralateral disease will remain eligible.
3. Tumor size < 1.5 cm in greatest diameter. Specifically, the tumor must measure < 1.5 cm in the axis parallel to the treatment probe and < 1.5 cm in the axis anti-parallel to the treatment probe. Largest size measured by required pre-treatment scans (mammogram, ultrasound and MRI) will be used to determine eligibility.
4. An ultrasound visible target for cryoablation:

   Ultrasound-visible mass or nonmass finding corresponding to the tumor or An ultrasound-visible biopsy marker placed within 1cm of the biopsied tumor.
5. No prior or planned neoadjuvant chemotherapy for breast cancer.
6. Adequate breast size for safe cryoablation. This will be determined by the interventional radiologist using a combination of clinical exam and imaging. Site of target for cryoablation must be greater than 1 cm from the nipple and greater than 1cm from the closest skin surface.

Exclusion Criteria:

1. Multifocal of multicentric carcinoma.
2. Pre-registration core biopsy with diagnosis of frank invasive carcinoma (not microinvasion) or lobular carcinoma.
3. Prior or planned neoadjuvant chemotherapy for breast cancer.
4. Retroglandular breast implants. (Please note that patients with retropectoral implants are allowed to enroll if they meet all other inclusion criteria.)

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
complete tumor ablation | 2 years
  rate of complete tumor ablation defined as no remaining invasive or in situ carcinoma present upon pathological examination of excised tissue

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Plaza, MD, Principal Investigator — Diagnostic Center for Women; Ahkeel Allen, MD, Principal Investigator — Breast Care Center Miami
Locations (2):
- United States (2):
  - Breast Care Center Miami, Miami, Florida
  - Diagnostic Center for Women, Miami, Florida